CLINICAL TRIAL: NCT01133405
Title: Single-Ascending Dose, Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study of LY2886721 in Healthy Subjects
Brief Title: A Safety Study of LY2886721 Single Doses in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 13733; I4O-MC-BACA (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-05

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — N-(3-(2-amino-4a,5,7,7a-tetrahydro-4H-furo(3,4-d)(1,3)thiazin-7a-yl)-4-fluorophenyl)-5-fluoropicolinamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- LY2886721 Part 1: Cohort A/B (Experimental): Single (7 milligram (mg), 15 mg, 25 mg, 35 mg) doses of LY2886721 administered orally in up to three of three study periods
  Interventions: Drug: LY2886721
- Placebo Part 1: Cohort A/B (Placebo Comparator): Single dose in up to 1 period
  Interventions: Drug: Placebo
- LY2886721 Part 2: Cohort C (Experimental): Single 10 mg dose of LY2886721, dose determined by Part 1
  Interventions: Drug: LY2886721
- LY2886721 Part 2: Cohort D (Experimental): Single 35 mg dose of LY2886721, dose determined by Part 1
  Interventions: Drug: LY2886721
- Placebo Part 2: Cohort C/D (Placebo Comparator): Single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2886721 — Oral capsules
  Arms: LY2886721 Part 1: Cohort A/B; LY2886721 Part 2: Cohort C; LY2886721 Part 2: Cohort D
Drug: Placebo — Oral capsules
  Arms: Placebo Part 1: Cohort A/B; Placebo Part 2: Cohort C/D

SUMMARY:
This is a Phase 1 study in healthy subjects to evaluate the safety and tolerability of LY2886721 single doses, how the body handles the drug, and the drug's effect on the body.

DETAILED DESCRIPTION:
This is a Phase 1 study with 2 parts, both in healthy subjects. Part 1 is a subject- and investigator-blind, placebo-controlled, randomized, 3-period, crossover study. Part 1 will assess the safety and tolerability of LY2886721 single doses, how the body handles the drug, and the drug's effect on the body. Part 2 is a subject- and investigator-blind, placebo-controlled, randomized study to assess the safety and tolerability of an LY2886721 single dose, how the body handles the drug, and the drug's effect on the body including in cerebrospinal fluid.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and nonchild-bearing potential women
* 20 years or older
* Body mass index between 18-32 kilograms per square meter (kg/m^2)

Exclusion Criteria:

* Taking over-the-counter or prescription medication with the exception of vitamins or minerals or stable doses of thyroid or estrogen hormone replacement
* Smoke more than 10 cigarettes per day

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beverly Hills, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consists of 2-parts. Part A was a cross-over study and was conducted in 2 alternating cohorts (Cohorts A and B). Part B was a single-dose, single period study in 2 cohorts (Cohorts C and D). All doses were administered in the fasted state, unless otherwise indicated. Each oral dose was followed by a washout period of at least 14 days.
Groups:
- Cohort A (Part 1) : Sequence 1: Participants received Placebo, 15 milligram (mg) LY2886721 and 35 mg LY2886721 orally as per the below dosing sequence in each period.
  Period 1: Placebo, Period 2: 15 mg LY2886721 and Period 3: 35 mg LY2886721.
- Cohort A (Part 1): Sequence 2: Participants received 1 mg LY2886721, 15 mg LY2886721 and placebo orally as per the below dosing sequence in each period.
  Period 1: 1 mg LY2886721, Period 2: 15 mg LY2886721 and Period 3: Placebo.
- Cohort A (Part 1): Sequence 3: Participants received 1 mg LY2886721, placebo and 35 mg LY2886721 orally as per the below dosing sequence in each period.
  Period 1: 1 mg LY2886721, Period 2: Placebo and Period 3: 35 mg LY2886721.
- Cohort B (Part 1): Sequence 1: Participants received 7 mg LY2886721, 25 mg LY2886721 and placebo and orally as per the below dosing sequence in each period.
  Period 1: 7 mg LY2886721, Period 2: 25 mg LY2886721 and Period 3: Placebo.
- Cohort B (Part 1): Sequence 2: Participants received 7 mg LY2886721, placebo and 7 mg LY2886721 (fed state) orally as per the below dosing sequence in each period.
  Period 1: 7 mg LY2886721 Period 2: Placebo and Period 3: 7 mg LY2886721 (fed state).
- Cohort B (Part 1): Sequence 3: Participants received Placebo, 25 mg LY2886721 and 7 mg LY2886721 (fed state) orally as per the below dosing sequence in each period.
  Period 1: Placebo, Period 2: 25 mg LY2886721 and Period 3: 7 mg LY2886721 (fed state).
- Cohort C (Part 2): 10mg LY2886721: Participants received a single 10 mg LY2886721 oral dose (low dose) in the fasted state.
- Cohort C (Part 2): Placebo; Cohort D (Part 2): Placebo: Participants received a single oral placebo dose in the fasted state.
- Cohort D (Part 2): 35 mg LY2886721: Participants received a single 35 mg LY2886721 oral dose (high dose) in the fasted state.
Period: Period 1
Arm/Group | Cohort A (Part 1) : Sequence 1 | Cohort A (Part 1): Sequence 2 | Cohort A (Part 1): Sequence 3 | Cohort B (Part 1): Sequence 1 | Cohort B (Part 1): Sequence 2 | Cohort B (Part 1): Sequence 3 | Cohort C (Part 2): 10mg LY2886721 | Cohort C (Part 2): Placebo | Cohort D (Part 2): 35 mg LY2886721 | Cohort D (Part 2): Placebo
Started | 3 | 6 | 5 | 5 | 3 | 5 | 5 | 2 | 4 | 2
Safety Analysis Population | 2 (One discontinued from study after randomization but before any study procedures.) | 6 | 5 | 5 | 3 | 5 | 5 | 2 | 4 | 2
Received at Least 1 Dose of Drug | 2 | 4 | 4 | 3 | 3 | 4 | 4 | 2 | 4 | 2
Completed | 2 | 3 | 4 | 1 | 3 | 3 | 4 | 2 | 4 | 2
Not Completed | 1 | 3 | 1 | 4 | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Discontinued after randomization | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Received drug only in period 2 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Received drug only in period 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Cohort A (Part 1) : Sequence 1 | Cohort A (Part 1): Sequence 2 | Cohort A (Part 1): Sequence 3 | Cohort B (Part 1): Sequence 1 | Cohort B (Part 1): Sequence 2 | Cohort B (Part 1): Sequence 3 | Cohort C (Part 2): 10mg LY2886721 | Cohort C (Part 2): Placebo | Cohort D (Part 2): 35 mg LY2886721 | Cohort D (Part 2): Placebo
Started | 2 | 4 (One participant started and received 15 mg LY2886721 only in period 2.) | 4 | 3 (Two participants started and received 25 mg LY2886721 only in period 2.) | 3 | 4 (One participant started and received 25 mg LY2886721 only in period 2.) | 0 (Cohort C was planned only for single period.) | 0 (Cohort C was planned only for single period.) | 0 (Cohort D was planned only for single period.) | 0 (Cohort D was planned only for single period.)
Received at Least 1 Dose of Study Drug | 2 | 4 | 4 | 3 | 3 | 4 | 0 | 0 | 0 | 0
Completed | 2 | 3 | 3 | 2 | 3 | 2 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Entry Criteria Not Met | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Cohort A (Part 1) : Sequence 1 | Cohort A (Part 1): Sequence 2 | Cohort A (Part 1): Sequence 3 | Cohort B (Part 1): Sequence 1 | Cohort B (Part 1): Sequence 2 | Cohort B (Part 1): Sequence 3 | Cohort C (Part 2): 10mg LY2886721 | Cohort C (Part 2): Placebo | Cohort D (Part 2): 35 mg LY2886721 | Cohort D (Part 2): Placebo
Started | 2 | 4 (One participant started and received placebo only in period 3.) | 4 (One participant started and received 35 mg LY2886721 only in period 3.) | 2 | 3 | 2 | 0 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug | 2 | 4 | 4 | 2 | 3 | 2 | 0 | 0 | 0 | 0
Completed | 2 | 4 | 4 | 2 | 3 | 2 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis population
Groups:
- Cohort A (Part 1): Sequence 1: Participants received Placebo, 15 milligram (mg) LY2886721 and 35 mg LY2886721 orally as per the dosing sequence in each period.
- Cohort A (Part 1): Sequence 2: Participants received 1 mg LY2886721, 15 mg LY2886721 and placebo orally as per the dosing sequence in each period.
- Cohort A (Part 1): Sequence 3: Participants received 1 mg LY2886721, placebo and 35 mg LY2886721 orally as per the dosing sequence in each period.
- Cohort B (Part 1): Sequence 1: Participants received 7 mg LY2886721, 25 mg LY2886721 and placebo and orally as per the dosing sequence in each period.
- Cohort B (Part 1): Sequence 2: Participants received 7 mg LY2886721, placebo and 7 mg LY2886721 (fed state) orally as per the dosing sequence in each period.
- Cohort B (Part 1): Sequence 3: Participants received Placebo, 25 mg LY2886721 and 7 mg LY2886721 (fed state) orally as per the below dosing sequence in each period.
- Cohort C (Part 2): Placebo: .Participants received a single oral placebo dose in the fasted state.
- Total: Total of all reporting groups
Arm/Group | Cohort A (Part 1): Sequence 1 | Cohort A (Part 1): Sequence 2 | Cohort A (Part 1): Sequence 3 | Cohort B (Part 1): Sequence 1 | Cohort B (Part 1): Sequence 2 | Cohort B (Part 1): Sequence 3 | Cohort C (Part 2): 10mg LY2886721 | Cohort C (Part 2): Placebo | Cohort D (Part 2): 35 mg LY2886721 | Cohort D (Part 2): Placebo | Total
Number analyzed (Participants) | 2 | 6 | 5 | 5 | 3 | 5 | 5 | 2 | 4 | 2 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 6 | 5 | 5 | 3 | 5 | 5 | 2 | 4 | 2 | 39
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 3 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 7
  Male | 2 | 6 | 2 | 5 | 1 | 5 | 4 | 1 | 4 | 2 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Asian | 1 | 3 | 1 | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 1 | 0 | 2 | 4 | 2 | 1 | 1 | 13
  White | 1 | 1 | 3 | 0 | 2 | 0 | 1 | 0 | 2 | 1 | 11
  More than one race | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 6 | 5 | 5 | 3 | 5 | 5 | 2 | 4 | 2 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Effects (Adverse Events)
Description: A summary of serious adverse events and other nonserious adverse events located in Reported Adverse Event section. To assess effect of food on pharmacokinetics of LY2886721, participants in Cohort B during Period 3 (1 period=8 days) of Part 1 fasted overnight for at least 8 hours prior to receiving a single 7-milligram (mg) oral dose of LY2886721 in the fed state (Part 1 - Fed). Participants in other LY2886721 groups received LY2886721 in fasted state. Due to crossover design in Part 1, results reported by treatment; thus, participants are included in multiple arms.
Time Frame: Predose to 10-14 days after final dose of study drug (up to 42 days)
Population: 39 of the 40 participants who were entered and randomized into the study and who had undergone study procedures were included in the safety analyses. One participant, who was entered and randomized into the study but did not undergo study procedures, was excluded from the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo (Part 1): In a single 8-day period, participants received a single placebo oral dose after an overnight fast.
- 1 mg LY2886721 (Part 1): In a single 8-day period, participants received a single 1-mg LY2886721 oral dose after an overnight fast.
- 7 mg LY2886721 (Part 1 - Fed and Fasted): In a single 8-day period, participants received a single 7-mg LY2886721 oral dose after an overnight fast, but 15 minutes after completing breakfast (Fed).
  In a single 8-day period, participants received a single 7-mg LY2886721 oral dose after an overnight fast (Fasted).
- 10 mg LY2886721 (Part 2): Participants received a single 10-mg LY2886721 oral dose after an overnight fast.
- 15 mg LY2886721 (Part 1): In a single 8-day period, participants received a single 15-mg LY2886721 oral dose after an overnight fast.
- 25 mg LY2886721 (Part 1): In a single 8-day period, participants received a single 25-mg LY2886721 oral dose after an overnight fast.
- 35 mg LY2886721 (Part 1): In a single 8-day period, participants received a single 35-mg LY2886721 oral dose after an overnight fast.
- 35 mg LY2886721 (Part 2): Participants received a single 35-mg LY2886721 oral dose after an overnight fast.
- Placebo (Part 2): Participants received a single placebo oral dose after an overnight fast.
Arm/Group | Placebo (Part 1) | 1 mg LY2886721 (Part 1) | 7 mg LY2886721 (Part 1 - Fed and Fasted) | 10 mg LY2886721 (Part 2) | 15 mg LY2886721 (Part 1) | 25 mg LY2886721 (Part 1) | 35 mg LY2886721 (Part 1) | 35 mg LY2886721 (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 19 | 8 | 8 | 4 | 6 | 7 | 6 | 4 | 4
Participants
  Serious Adverse Events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other Nonserious Adverse Events | 4 | 2 | 1 | 1 | 0 | 1 | 3 | 4 | 3

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of LY2886721
Description: To assess effect of food on pharmacokinetics of LY2886721, participants in Cohort B during Period 3 (1 period=8 days) of Part 1 fasted overnight for at least 8 hours prior to receiving a single 7-milligram (mg) oral dose of LY2886721 in the fed state (Part 1 - Fed). Participants in the other LY2886721 groups received LY2886721 in the fasted state. Due to the crossover design in Part 1, results are reported by treatment; therefore, participants are included in multiple arms.
Time Frame: 0, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60 and 96 hours post-dose
Population: All participants who received at least 1 dose of LY2886721 and have evaluable pharmacokinetic data were included in the analysis. One participant from Part 2, who experienced an adverse event before receiving study medication, was not included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- 7 mg LY2886721 Fed (Part 1): In a single 8-day period, participants received a single 7-mg LY2886721 oral dose after an overnight fast, but 15 minutes after completing breakfast.
- 7 mg LY2886721 Fasted (Part 1): In a single 8-day period, participants received a single 7-mg LY2886721 oral dose after an overnight fast.
Arm/Group | 1 mg LY2886721 (Part 1) | 7 mg LY2886721 Fed (Part 1) | 7 mg LY2886721 Fasted (Part 1) | 10 mg LY2886721 (Part 2) | 15 mg LY2886721 (Part 1) | 25 mg LY2886721 (Part 1) | 35 mg LY2886721 (Part 1) | 35 mg LY2886721 (Part 2)
Number analyzed (Participants) | 8 | 5 | 6 | 4 | 6 | 7 | 6 | 4
nanogram per milliliter (ng/mL) | 1.9 (65) | 22.5 (23) | 18.2 (64) | 6.6 (60) | 41.6 (24) | 79.1 (25) | 78.2 (45) | 53.3 (44)

3. Secondary Outcome: Plasma Concentration of LY2886721: Area Under the Concentration Versus Time Curve (AUC)
Description: Pharmacokinetic AUC for LY2886721 from time 0 to infinity. To assess effect of food on pharmacokinetics of LY2886721, participants in Cohort B during Period 3 (1 period=8 days) of Part 1 fasted overnight for at least 8 hours prior to receiving a single 7-milligram (mg) oral dose of LY2886721 in the fed state (Part 1 - Fed). Participants in the other LY2886721 groups received LY2886721 in the fasted state. Due to the crossover design in Part 1, results are reported by treatment; therefore, participants are included in multiple arms.
Time Frame: 0, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60 and 96 hours post-dose
Population: All participants who received at least 1 dose of LY2886721 and have evaluable pharmacokinetic data were included in the analysis. One participant in Part 2, who experienced an adverse event before receiving study medication, was not included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | 1 mg LY2886721 (Part 1) | 7 mg LY2886721 Fed (Part 1) | 7 mg LY2886721 Fasted (Part 1) | 10 mg LY2886721 (Part 2) | 15 mg LY2886721 (Part 1) | 25 mg LY2886721 (Part 1) | 35 mg LY2886721 (Part 1) | 35 mg LY2886721 (Part 2)
Number analyzed (Participants) | 8 | 5 | 6 | 4 | 6 | 7 | 6 | 4
nanogram*hour per milliliter (ng*h/mL) | NA (NA) — Data for the 1-mg LY2886721 group are not presented for this outcome measure because sufficient data did not exist for the terminal elimination phase calculations. | 311 (14) | 212 (41) | 144 (580) | 468 (20) | 926 (16) | 954 (37) | 800 (38)

4. Secondary Outcome: Pharmacodynamic Biomarker: Plasma Amyloid Beta (Aβ) 1-40 Concentration (Part 1 Only)
Description: Plasma concentrations of Aβ1-40 were based on the lowest observed/measured concentration (Cnadir). To assess effect of food on pharmacokinetics of LY2886721, participants in Cohort B during Period 3 (1 period=8 days) of Part 1 fasted overnight for at least 8 hours prior to receiving a single 7-milligram (mg) oral dose of LY2886721 in the fed state (Part 1 - Fed). Participants in the other LY2886721 groups received LY2886721 in the fasted state. Due to the crossover design in Part 1, results are reported by treatment; therefore, participants are included in multiple arms.
Time Frame: 0, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60 and 96 hours post-dose
Population: All participants who received at least 1 dose of LY2886721 in Part 1 and have evaluable pharmacodynamic data were included in the analysis. One participant who was entered and randomized into the study but did not undergo study procedures, was excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram per milliliter (pg/mL)
Arm/Group | Placebo (Part 1) | 1 mg LY2886721 (Part 1) | 7 mg LY2886721 (Part 1 - Fed and Fasted) | 15 mg LY2886721 (Part 1) | 25 mg LY2886721 (Part 1) | 35 mg LY2886721 (Part 1)
Number analyzed (Participants) | 19 | 8 | 6 | 6 | 7 | 6
picogram per milliliter (pg/mL) | 121 (23.6) | 80 (19.5) | 56 (41.3) | 35 (37.7) | 34 (28.4) | 36 (11.7)

5. Secondary Outcome: Cerebrospinal Fluid (CSF) Maximum Observed Drug Concentration (Cmax) of LY2886721 (Part 2 Only)
Time Frame: Predose and up to 36 hours postdose
Population: All participants who received at least 1 dose of LY2886721 in Part 2 and have evaluable pharmacokinetic data were included in the analysis. One participant, who experienced an adverse event before receiving study medication, was not included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- 35 mg LY2886721 (Part 2): Participants received a single 35-mg LY2886721 oral dose by mouth after an overnight fast.
Arm/Group | 10 mg LY2886721 (Part 2) | 35 mg LY2886721 (Part 2)
Number analyzed (Participants) | 4 | 4
nanogram per milliliter (ng/mL) | 0.93 (60) | 5.99 (39)

6. Secondary Outcome: Cerebrospinal Fluid (CSF) Pharmacodynamic Biomarker Amyloid Beta (Aβ) 1-40 Concentration (Part 2 Only)
Description: CSF Aβ 1-40 concentration was based on the lowest observed/measured concentration (Cnadir).
Time Frame: Predose and up to 36 hours postdose
Population: All participants who received at least 1 dose of LY2886721 in Part 2 and have evaluable pharmacodynamic data were included in the analysis. One participant, who experienced an adverse event before receiving study medication, was not included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram per milliliter (pg/mL)
Arm/Group | 10 mg LY2886721 (Part 2) | 35 mg LY2886721 (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 4 | 4 | 4
picogram per milliliter (pg/mL) | 8080 (48.8) | 5650 (51.1) | 7150 (62.4)

7. Secondary Outcome: Cerebrospinal Fluid (CSF) Area Under the Concentration Versus Time Curve (AUC) of LY2886721 (Part 2 Only)
Time Frame: Predose and up to 36 hours postdose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | 10 mg LY2886721 (Part 2) | 35 mg LY2886721 (Part 2)
Number analyzed (Participants) | 4 | 4
nanogram*hour per milliliter (ng*h/mL) | 27 (89) | 121 (30)

ADVERSE EVENTS:
Groups:
- 7 mg LY2886721 (Part 1 - Fed and Fasted): In a single 8-day period, participants received a single 7-mg LY2886721 oral dose after an overnight fast, but 15 minutes after breakfast (Fed).
  In a single 8-day period, participants received a single 7-mg LY2886721 oral dose after an overnight fast (Fasted).
Arm/Group | Placebo (Part 1) | 1 mg LY2886721 (Part 1) | 7 mg LY2886721 (Part 1 - Fed and Fasted) | 10 mg LY2886721 (Part 2) | 15 mg LY2886721 (Part 1) | 25 mg LY2886721 (Part 1) | 35 mg LY2886721 (Part 1) | 35 mg LY2886721 (Part 2) | Placebo (Part 2)
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/8 | 0/8 | 0/4 | 0/6 | 0/7 | 0/6 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/19 | 2/8 | 1/8 | 1/4 | 0/6 | 1/7 | 3/6 | 4/4 | 3/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part 1) (N=19) | 1 mg LY2886721 (Part 1) (N=8) | 7 mg LY2886721 (Part 1 - Fed and Fasted) (N=8) | 10 mg LY2886721 (Part 2) (N=4) | 15 mg LY2886721 (Part 1) (N=6) | 25 mg LY2886721 (Part 1) (N=7) | 35 mg LY2886721 (Part 1) (N=6) | 35 mg LY2886721 (Part 2) (N=4) | Placebo (Part 2) (N=4)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days